CLINICAL TRIAL: NCT05219045
Title: One-Year Impact Evaluation of Ohio Retaining Employment and Talent After Injury/Illness Network (RETAIN)
Brief Title: Ohio RETAIN Impact Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Social Security Administration (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RTN-OH
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-11

CONDITIONS: Disability
Keywords: disability; employment; unemployment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RETAIN Programming (Experimental): The experimental group receives the full set of RETAIN intervention activities.
  Interventions: Other: Ohio RETAIN
- Control (No Intervention): Medical providers who treat both treatment and control group enrollees receive training on stay-at-work/return-to-work best practices

INTERVENTIONS:
Other: Ohio RETAIN — RETAIN projects include a combination of medical provider services, stay-at-work/return-to-work (SAW/RTW) coordination services, and other SAW/RTW services. The evaluation compares the treatment group that is eligible to receive the full set of RETAIN intervention activities and an active comparator that is not.
  Arms: RETAIN Programming

SUMMARY:
The Retaining Employment and Talent after Injury/Illness Network (RETAIN) demonstration is a collaborative effort between the U.S. Department of Labor (DOL) and the Social Security Administration (SSA) to improve employment outcomes for individuals who experience injuries or illnesses that put them at risk of exiting the labor force and relying on disability programs and other public supports in the long term. RETAIN projects include a combination of medical provider services, stay-at-work/return-to-work (SAW/RTW) coordination services, and other SAW/RTW services. This evaluation will focus on the Ohio Department of Job and Family Services' implementation of "Ohio RETAIN." The evaluation will document how the project is implemented, describe enrollees, estimate the project's impacts on enrollees' outcomes, and assess whether the benefits outweigh the costs.

DETAILED DESCRIPTION:
The Ohio Department of Job and Family Services has partnered with Mercy Health to implement "Ohio RETAIN" in Youngstown, Toledo and Cicinnati catchment areas. SSA contracted with Mathematica to conduct an independent evaluation of the program.

Under the RETAIN model medical providers receive training and incentives to use occupational health best practices. The state agency also coordinates SAW/RTW services for the enrollee, fosters communication among Ohio RETAIN stakeholders about the treatment enrollee returning to work, and monitors the enrollee's medical and employment progress. The Business Resource Network and OhioMeansJobs provide additional support for workplace-based interventions and retaining or rehabilitation of enrollees.

Ohio recruits potentially eligible workers as they receive care from medical providers. The evaluation team randomly assigns each enrollee to either a treatment group that is eligible to receive the full set of RETAIN intervention activities or a control group that is not. The evaluation team then compares the outcomes of the treatment and control groups and gathers evidence on how Ohio RETAIN shaped the outcomes of enrollees who were eligible for its services, regardless of whether they participated in those services. Data sources include enrollment data, surveys, administrative records, program data, and qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 65
* Currently employed or actively seeking employment
* Live in Youngstown (Mahoning, Columbiana, and Trumbull Counties), Toledo (Lucas County), and Cincinnati (Butler, Clermont, Hamilton, and Warren Counties
* Provider prescribed limitations of work, FMLA paperwork submitted for provider completion, documentation of work limitations in office notes, or an illness/injury which has previously resulted in work limitations based upon the nurse's clinical judgement and experience for a treatment barrier that is prolonging recovery and return to work
* Has a qualifying musculoskeletal injury or exacerbation or a qualifying cardiovascular procedure

  * Qualifying musculoskeletal injury or exacerbation: (a) Has occurred in the last 3 months and has limited their ability to work; (b) Not work related; (c) Surgery was in the last 3 months with continued limitations at work; (d) Upcoming surgery within 1 month.
  * Qualifying Cardiovascular procedure: (a) CABG (Coronary Artery Bypass Graft) scheduled or done; (b) TAVR (Coronary Valve replacement with open heart entry to exclude trans-catheter) approach scheduled or done; (c) (Abdominal Aortic Aneurysm) open entry approach scheduled or done; (d) Aorto-bifemoral bypass with activity restrictions for 4 weeks or more scheduled or done; (e) Cardiac Catheterization with stent placement with: i) Cardiac Rehab ordered at time of Cardiac Catheterization or ii) No Cardiac Rehab ordered at time of Cardiac Catheterization, but Cardiac Rehab has been ordered at Cardiac Catheterization follow up appointment.

Exclusion Criteria:

* Retired
* Has or is pursuing a Bureau of Workers' Compensation claim for this injury
* Has applied for or is currently receiving Social Security Insurance or Social Security Disability Insurance
* Has substance abuse disorder
* Has legal representation
* Pregnant
* Has a terminal disease
* Multiple trauma patient with multi-system involvement requiring being off work/recovery for more than 3-6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3200 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Share of enrollees employed in the fourth quarter after enrollment | Measured over the three months in the fourth quarter after enrollment
  Share of enrollees employed in the fourth quarter after enrollment obtained from state unemployment insurance wage records. These files include individual-level wage records for six quarters surrounding enrollment in the study, including the quarter prior to enrollment, the quarter of enrollment, and four post-enrollment quarters.
Enrollee earnings in the fourth quarter after enrollment | Measured over the three months in the fourth quarter after enrollment
  Sum of enrollee earnings in the fourth quarter after enrollment obtained from state unemployment insurance wage records. These files include individual-level wage records for six quarters surrounding enrollment in the study, including the quarter prior to enrollment, the quarter of enrollment, and four post-enrollment quarters.
Share of enrollees that applied for SSDI or SSI during the 12 months after enrollment | Measured in the 12 months after enrollment
  Share of enrollees that applied for SSDI or SSI during any of the 12 months after enrollment obtained from SSA program data. These files include detailed information about Social Security Disability Insurance (SSDI) and Supplemental Security Income (SSI) applications SSDI and SSI awards, SSDI and SSI benefit amounts and enrollee characteristics (for enrollees who have ever applied for SSA program benefits)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Berk, PhD, Principal Investigator — Mathematica Policy Research, Inc.
Locations (1):
- Ohio Department of Job and Family Services (ODJFS), Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No